CLINICAL TRIAL: NCT00609596
Title: An Open Label, Randomized, Repeat Dose, 3 Period Crossover Study to Determine the Bioequivalence of 3 Different Formulations of Tamsulosin at Steady State in Healthy Male Volunteers
Brief Title: A Study To Compare 3 Different Formulations Of Tamsulosin At Steady State.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ARI111402
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Prostatic Hyperplasia
Keywords: dutasteride; tamsulosin; benign prostatic hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: GI198745

INTERVENTIONS:
Drug: GI198745

SUMMARY:
Dutasteride and tamsulosin are to treat benign prostatic hyperplasia. Studies show that when given together, there is more improvement in symptoms than either drug alone. In this study, we are looking to see if 2 different formulations of tamsulosin in our combination capsules are the same after 7 days of dosing as the US commercial tamsulosin and dutasteride.

ELIGIBILITY:
Inclusion criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with orthostasis at screening should be excluded from enrollment.
* Males between 18 and 45 years of age (inclusive).
* Male subjects must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study medication until follow-up from the study.
* Body weight </ 55 kg and BMI within the range 19.0 - 30.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF < 450 msec.
* Subjects must agree not to donate blood and blood products for 6 months after the last dose of study medication.

Exclusion criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Slow metabolizer for CYP2D6 as determined by screening PGx analysis.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:

  - An average weekly intake of >14 drinks/week. One drink is equivalent to: 12 g alcohol = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication and until collection of the final PK sample from the study, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof, including sulfonamides, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of postural hypotension, dizziness, poor hydration, vertigo, vaso-vagal reactions or any other signs and symptoms of orthostasis, which in the opinion of the investigator could be exacerbated by tamsulosin and result in putting the subject at risk of injury.
* Orthostatic hypotension at screening, defined as a reduction in systolic blood pressure of 20 mmHg or more and/or a reduction in diastolic blood pressure of 10 mmHg or more for standing vs. supine measurements.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Consumption of red wine, seville oranges, grapefruit, grapefruit juice or cruciferous vegetables (watercress, broccoli, cabbage, Brussels sprouts) from 7 days prior to the first dose of study medication and until collection of the final PK sample in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02-26 (Actual); Primary Completion 2008-04-23 (Actual); Study Completion 2008-04-23 (Actual)

PRIMARY OUTCOMES:
PK at 0,1,2,3,4,5,6,7,8,10,12,16,24,36,48,72

SECONDARY OUTCOMES:
Clinical safety labs | at check in
measurement of orthostatic hypotension | at 6 hours post dose on days 1 and 7
adverse event reporting
C(tau) (pre-dose concentrations determined immediately before a dose at steady state), t1/2, tmax, lambda, Cmin and fluctuation [(Cmax - Cmin)/(AUC(0-24)/24)] of tamsulosin, as data permit.
Safety and tolerability of all treatments as assessed by blood pressure and pulse rate measurements, adverse events and clinical laboratory safety tests.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Cai G, Thiessen JJ, Baidoo CA, Fossler MJ. Operating characteristics of a partial-block randomized crossover bioequivalence study for dutasteride, a drug with a long half-life: investigation through simulation and comparison with final results. J Clin Pharmacol. 2010 Oct;50(10):1142-50. doi: 10.1177/0091270009355155. Epub 2010 Feb 16. PMID 20160156
- See also: Results for study ARI111402 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/ARI111402?search=study&study_ids=ARI111402#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: ARI111402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ARI111402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ARI111402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: ARI111402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ARI111402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ARI111402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ARI111402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register